CLINICAL TRIAL: NCT02026180
Title: Randomized Comparison of Micropuncture vs. Standard Common Femoral Artery Access for Reducing Vascular Access Complications
Brief Title: Micropuncture vs. Standard Common Femoral Artery Access
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low incidence of primary endpoint
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, MD, PhD, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-090
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Vascular Access Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropuncture Access (Active Comparator): Vascular access using micropuncture needle kit
  Interventions: Device: Micropuncture Access
- Standard 18G vascular access needle (Active Comparator): Vascular access using standard 18G needle
  Interventions: Device: Micropuncture Access

INTERVENTIONS:
Device: Micropuncture Access — Femoral arterial access will be obtained either with a 21G micropuncture needle kit or an 18G standard access needle.

SUMMARY:
Vascular access complications can occur during or after cardiac or peripheral arterial catheterization. These complications increase patient morbidity and mortality, as well as healthcare costs. Several strategies and devices have been employed to decrease the risk for vascular access complications, such as fluoroscopy-guided access, ultrasound-guided access and vascular closure devices. Randomized trial data has failed to demonstrate that fluoroscopic guidance reduces common femoral artery access complications. While meta-analysis data has demonstrated that vascular closure devices decrease time to arterial hemostasis, increase patient mobilization and facilitate earlier patient discharge, they do not reduce the incidence of vascular complications as compared to hemostasis achieved with manual pressure. Ultrasound guidance has been shown to facilitate femoral artery access and reduce femoral artery vascular complications. A new device, the Micropuncture Kit (Cook Medical, Bloomington, IN) allows vascular access with a small 21gauge needle as opposed to the standard method, which requires an 18 gauge needle. The use of the Micropuncture Kit for the purpose of decreasing vascular access complications has not been examined in a randomized study to date.

The present study is a 552 patient randomized controlled clinical trial that will help determine whether femoral arterial access obtained using the Micropuncture Kit will reduce the incidence of vascular access complications compared to the standard 18 gauge needle.

The specific aim of this proposal is to compare the rate of femoral artery access complications using the Micropuncture Kit vs. standard femoral artery access.

It is our hypothesis that the incidence of femoral artery access complications will be lower among patients in whom the Micropuncture Kit is used.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing left heart or peripheral catheterization through the common femoral artery with anticipated or possible percutaneous coronary or peripheral intervention

Exclusion Criteria:

1. Arterial access obtained through the radial or brachial artery
2. Age less than 18 years
3. Patients with known bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Arterial perforation | 30 days
Acute limb ischemia | 30 days
  Acute limb ischemia, indicated by thrombosis or loss of distal pulses
Arteriovenous fistula | 30 days
  Arteriovenous fistula, defined as an abnormal communication between an artery and a vein
Access site pseudoaneurysm | 30 days
Retroperitoneal bleeding | 30 days
  Retroperitoneal bleeding defined as computerized tomography confirmation of femoral artery hemorrhage into the retroperitoneal space
Groin hematoma | 30 days
  Groin hematoma, defined as hematoma >5 cm.
Femoral artery dissection | 30 days
  Femoral artery dissection confirmed by angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States